CLINICAL TRIAL: NCT07071675
Title: Postoperative Pain and Flare-Up Incidence Following the Use of Bio Ceramic Based Intra-Canal Medication in Diabetic Type II Patients (A Randomized Clinical Trial)
Brief Title: Postoperative Pain and Flare-Up Rates in Diabetic Type II Patients Following The Use of Bioceramic Intracanal Medication
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abdulrahman Issam Abdulkareem Marie, Postgraduate Student, Department of Endodontics, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-EC Research NO.1064
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Flare Up, Symptom; Flare up; Diabete Type 2
Keywords: postoperative pain; flare up; diabetes type II; Intra-Canal medication; bioceramic; calcium hydroxide
MeSH Terms: conditions — Pain, Postoperative; Symptom Flare Up; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. Each group will receive a different intracanal medicament following root canal treatment. Postoperative pain and flare-up incidence will be assessed and compared between the two groups.
Who Masked: Participant
Masking Description: Participants will be blinded to the type of intracanal medicament used during their root canal treatment. The medicaments will be applied in a manner that prevents participants from identifying which treatment they received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium Hydroxide Group (GROUP I) (Experimental): Treated using calcium hydroxide as an intracanal medicament (n=28)
  Interventions: Drug: Calcium Hydroxide Intracanal medication
- Bioceramic Group (GROUP II) (Experimental): treated using bio-ceramic based material as an intracanal medicament (n=28)
  Interventions: Drug: bioceramic based intracanal medication

INTERVENTIONS:
Drug: Calcium Hydroxide Intracanal medication — Treated using calcium hydroxide based material as an intracanal medicament
  Arms: Calcium Hydroxide Group (GROUP I)
Drug: bioceramic based intracanal medication — treated using bio-ceramic based material as an intracanal medicament
  Arms: Bioceramic Group (GROUP II)

SUMMARY:
The goal of this randomized clinical trial is to evaluate the Postoperative Pain and Flare-Up incidence following the use of Bio-Ceramic Based Intra-Canal Medication in Diabetic type II Patients compared to the Calcium Hydroxide based Intra-canal medicament.

The main questions it aims to answer are:

1. Is there any difference between using the two intracanal medicaments in the aspects of postoperative pain and flare-up incidence in diabetic type II patients?
2. Do intracanal medications reduce postoperative pain and flare-up incidence in diabetic type II patients?

Participants will be divided into two groups:

( both groups will receive root canal treatment in single rooted teeth) then: First group: will receive "Calcium Hydroxide based" intracanal medicament Second group: will receive "Bio-Ceramic Based" intracanal medicament

Postoperative pain will be assessed using:

* visual analog scale (VAS), A scale from (0 to 10) where "0" means no pain and "10" means a severe pain that has never faced before.
* Patients will be contacted by phone at 6, 12, 24, 48, 72 hours and 7 days after the first visit to collect the postoperative pain data.

Flare-up is assessed:

- by asking the patient to notify the investigator if any sudden severe pain or swelling takes place.

ELIGIBILITY:
Inclusion Criteria:

* Patients with controlled diabetes mellitus type II.
* Necrotic single rooted teeth:

  * with periapical lesion ranging (1-2mm) in diameter.
  * with complete root formation.
  * Without calcified root canals.
  * Without root caries.
  * Without external or internal root resorption.
  * Without anatomical abnormalities such as fusion.

Exclusion Criteria:

* Pregnant females.
* Patients with other systemic diseases in combination with diabetes mellitus.
* Patients under antibiotic or analgesic administration.
* Patients with facial swelling.
* Teeth that are not indicated for endodontic treatment: bad oral hygiene, mobile teeth, or recessed teeth.
* Previously endodontically treated teeth.
* Teeth with sinus tract.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
postoperative pain intensity | 6, 12, 24, 48, 72 hours and 7 days after the first visit to collect the postoperative pain data.
  Postoperative pain is to be assessed using visual analog scale (VAS), A scale from (0 to 10) where "0" means no pain and "10" means a severe pain that has never faced before.
  Patients will be contacted by phone at 6, 12, 24, 48, 72 hours and 7 days after the first visit to collect the postoperative pain data.
Flare-Up Incidence | Within 7 days post-treatment
  Flare-up is assessed through asking the patient to notify the investigator if any sudden severe pain or swelling takes place.
  This could require an unscheduled emergency visit or prescription of additional medication.

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to privacy concerns and the limited scope of data use approved by the ethics committee. The study is designed for internal analysis only and does not include provisions for public data sharing.